CLINICAL TRIAL: NCT07308314
Title: Taining Golden Lake Comprehensive Chronic Disease Management Initiative
Acronym: TAIGOLD-CDM
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Dajun Chai, Professor and Chief Physician, Department of Cardiology, First Affiliated Hospital of Fujian Medical University
Other Study IDs: MRCTA,ECFAH of FMU[2025]950
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-07

CONDITIONS: Chronic Disease; Chronic Disease Management; Hypertension; Diabetes Mellitus; Dyslipidemias; Frailty; Sarcopenia
Keywords: Chronic Disease Management; Prospective Cohort; Hypertension; Diabetes Mellitus; Dyslipidemia; Cardiovascular Disease; Frailty; Sarcopenia; Aging; Healthy Aging
MeSH Terms: conditions — Chronic Disease; Hypertension; Diabetes Mellitus; Dyslipidemias; Frailty; Sarcopenia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 15 mL fasting venous blood collected in the morning after an overnight fast. Used for routine hematology, biochemistry, platelet aggregation, BNP, CRP, and bone turnover markers. Aliquots will also be stored for future analyses. All biospecimens will be processed and stored according to standardized operating procedures. A biobank will be established at the county hospital and collaborating institutions to support future multi-omics and public health research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Taining County Resident Cohort: A community-based cohort of ≥20,000 adult residents (aged 18 years and older) living in Taining County, Fujian Province, China. Participants will undergo baseline assessments including questionnaires, physical examinations, laboratory tests, imaging, and biospecimen collection. Annual follow-up (active and passive) will be conducted for 3 years to record incidence of chronic diseases, functional status, and aging-related outcomes.

SUMMARY:
This study aims to establish the first county-level, population-based prospective cohort in Taining County, Fujian Province, China. The cohort will include at least 20,000 residents aged 18 years or older. The project will systematically collect questionnaires, physical measurements, laboratory tests, imaging data, and biological samples to build a multi-dimensional health database and biobank. Through 3-year follow-up, the study seeks to reveal the epidemiological patterns and risk factors of chronic diseases, characterize the natural course of multimorbidity and aging syndromes, and develop a comprehensive chronic disease management model suitable for rural and mountainous regions.

DETAILED DESCRIPTION:
China is undergoing rapid population aging, with chronic non-communicable diseases (NCDs) becoming the leading cause of death and disability. Taining County, located in a mountainous area of Fujian Province, faces a higher-than-average aging population and a growing burden of hypertension, diabetes, dyslipidemia, and cardiovascular diseases. Early detection and standardized management remain insufficient, and healthcare resources are limited. This study will establish a prospective cohort covering ≥20,000 residents, integrating demographic, lifestyle, clinical, laboratory, and imaging data. Active follow-up will be conducted annually, complemented by passive follow-up through local healthcare and death registry systems. The study will (1) identify epidemiological features and risk factors of common chronic diseases, (2) explore multimorbidity and aging trajectories, and (3) develop a replicable "Taining Model" for chronic disease prevention and management at the county level. The results will provide an evidence base for public health decision-making and chronic disease control strategies in similar rural and mountainous regions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female.
* Resident of Taining County for ≥6 months and expected to remain in the county for at least the next 3 years.
* Full civil capacity and able to understand study procedures.
* Willing to voluntarily participate and provide written informed consent.
* Able to complete baseline survey and follow-up visits.

Exclusion Criteria:

* Refusal to sign informed consent.
* Severe psychiatric disorders or cognitive impairment preventing participation.
* End-stage disease with expected survival <1 year.
* Long-term migrants (≥6 months per year outside the county), unable to guarantee follow-up.
* Participation in other clinical studies that may interfere with this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of community-dwelling adult residents of Taining County, a mountainous region in Fujian Province, China. Eligible participants are men and women aged 18 years and older who have lived in the county for at least 6 months and are expected to remain for the next 3 years.
  A total of at least 20,000 participants will be enrolled at baseline through community-based recruitment and household registration systems. The population reflects the demographic and health characteristics of a rural county with a relatively high proportion of older adults and a growing burden of chronic diseases such as hypertension, diabetes, and cardiovascular disease.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | Up to 36 months
  Composite outcome including cardiovascular death, non-fatal myocardial infarction, and non-fatal stroke. Events will be ascertained through active follow-up and confirmed using medical records and hospital discharge summaries.

SECONDARY OUTCOMES:
Incidence of Cardiovascular and Cerebrovascular Events | Up to 36 months
  New onset of coronary heart disease, stroke, or heart failure, identified through follow-up visits and confirmed using medical records.
Heart Failure-Related Rehospitalization Rate | Up to 36 months
  Rehospitalization due to worsening heart failure among participants diagnosed with heart failure, confirmed by hospital admission records.
Bleeding Events | Up to 36 months
  Occurrence of clinically significant bleeding events, including gastrointestinal bleeding and other major or clinically relevant non-major bleeding, identified through follow-up and medical records.
Health Economics Outcomes | Up to 36 months
  Direct medical costs, hospitalization expenses, outpatient visit costs, medication costs, and health service utilization related to chronic disease management, collected from medical records and insurance data.
Cognitive Function Outcomes | Baseline and annual follow-up (Year 1-3)
  Changes in cognitive function assessed using standardized cognitive screening tools administered at baseline and during follow-up.
Cancer Incidence and Cancer-Related Outcomes | Up to 36 months
  Newly diagnosed malignant tumors and cancer-related outcomes, identified through self-report and confirmed by medical records or cancer registry data.
All-Cause Mortality | Up to 36 months
  Death from any cause, confirmed through medical records and the local death registry system.

CONTACTS AND LOCATIONS:
Overall Officials: Dajun Chai, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including demographic information, clinical characteristics, imaging parameters ECG data, laboratory test results, biospecimen profiles and follow-up outcomes, will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available beginning 24 months after the primary study completion date and remain accessible for up to 24 months.
Access Criteria: Qualified researchers with a scientifically sound proposal may request access to the data. Requests will be evaluated by the study steering committee. Approved users must sign a data use agreement ensuring compliance with privacy, ethical, and scientific standards.
URL: https://www.fjmu.edu.cn

REFERENCES:
- [Background] Chen L, Li X, Lv Y, Tan X, Zhong VW, Rong S, Liu G, Liu L. Physical frailty, adherence to ideal cardiovascular health and risk of cardiovascular disease: a prospective cohort study. Age Ageing. 2023 Jan 8;52(1):afac311. doi: 10.1093/ageing/afac311. PMID 36626327
- [Background] Hu L, Li J, Tang Z, Gong P, Chang Z, Yang C, Ma T, Jiang S, Yang C, Zhang T. How does biological age acceleration mediate the associations of obesity with cardiovascular disease? Evidence from international multi-cohort studies. Cardiovasc Diabetol. 2025 May 14;24(1):209. doi: 10.1186/s12933-025-02770-0. PMID 40369582
- [Background] Global Cardiovascular Risk Consortium; Magnussen C, Ojeda FM, Leong DP, Alegre-Diaz J, Amouyel P, Aviles-Santa L, De Bacquer D, Ballantyne CM, Bernabe-Ortiz A, Bobak M, Brenner H, Carrillo-Larco RM, de Lemos J, Dobson A, Dorr M, Donfrancesco C, Drygas W, Dullaart RP, Engstrom G, Ferrario MM, Ferrieres J, de Gaetano G, Goldbourt U, Gonzalez C, Grassi G, Hodge AM, Hveem K, Iacoviello L, Ikram MK, Irazola V, Jobe M, Jousilahti P, Kaleebu P, Kavousi M, Kee F, Khalili D, Koenig W, Kontsevaya A, Kuulasmaa K, Lackner KJ, Leistner DM, Lind L, Linneberg A, Lorenz T, Lyngbakken MN, Malekzadeh R, Malyutina S, Mathiesen EB, Melander O, Metspalu A, Miranda JJ, Moitry M, Mugisha J, Nalini M, Nambi V, Ninomiya T, Oppermann K, d'Orsi E, Pajak A, Palmieri L, Panagiotakos D, Perianayagam A, Peters A, Poustchi H, Prentice AM, Prescott E, Riserus U, Salomaa V, Sans S, Sakata S, Schottker B, Schutte AE, Sepanlou SG, Sharma SK, Shaw JE, Simons LA, Soderberg S, Tamosiunas A, Thorand B, Tunstall-Pedoe H, Twerenbold R, Vanuzzo D, Veronesi G, Waibel J, Wannamethee SG, Watanabe M, Wild PS, Yao Y, Zeng Y, Ziegler A, Blankenberg S. Global Effect of Modifiable Risk Factors on Cardiovascular Disease and Mortality. N Engl J Med. 2023 Oct 5;389(14):1273-1285. doi: 10.1056/NEJMoa2206916. Epub 2023 Aug 26. PMID 37632466
- [Background] Moturi S, Ghosh-Choudhary SK, Finkel T. Cardiovascular disease and the biology of aging. J Mol Cell Cardiol. 2022 Jun;167:109-117. doi: 10.1016/j.yjmcc.2022.04.005. Epub 2022 Apr 11. PMID 35421400
- [Background] Liberale L, Badimon L, Montecucco F, Luscher TF, Libby P, Camici GG. Inflammation, Aging, and Cardiovascular Disease: JACC Review Topic of the Week. J Am Coll Cardiol. 2022 Mar 1;79(8):837-847. doi: 10.1016/j.jacc.2021.12.017. PMID 35210039
- [Background] Hu C. Prevention of cardiovascular disease for healthy aging and longevity: A new scoring system and related "mechanisms-hallmarks-biomarkers". Ageing Res Rev. 2025 May;107:102727. doi: 10.1016/j.arr.2025.102727. Epub 2025 Mar 15. PMID 40096912
- [Background] da Silva PFL, Schumacher B. Principles of the Molecular and Cellular Mechanisms of Aging. J Invest Dermatol. 2021 Apr;141(4S):951-960. doi: 10.1016/j.jid.2020.11.018. Epub 2021 Jan 29. PMID 33518357
- [Background] Moqri M, Herzog C, Poganik JR; Biomarkers of Aging Consortium; Justice J, Belsky DW, Higgins-Chen A, Moskalev A, Fuellen G, Cohen AA, Bautmans I, Widschwendter M, Ding J, Fleming A, Mannick J, Han JJ, Zhavoronkov A, Barzilai N, Kaeberlein M, Cummings S, Kennedy BK, Ferrucci L, Horvath S, Verdin E, Maier AB, Snyder MP, Sebastiano V, Gladyshev VN. Biomarkers of aging for the identification and evaluation of longevity interventions. Cell. 2023 Aug 31;186(18):3758-3775. doi: 10.1016/j.cell.2023.08.003. PMID 37657418
- [Background] Nash DB. The Future of Chronic Disease Management. Popul Health Manag. 2023 Aug;26(S1):S2-S3. doi: 10.1089/pop.2023.0128. No abstract available. PMID 37603800
- [Background] Elendu C, Elendu RC, Enyong JM, Ibhiedu JO, Ishola IV, Egbunu EO, Meribole ES, Lawal SO, Okenwa CJ, Okafor GC, Umeh ED, Mutalib OO, Opashola KA, Fatoye JO, Awotoye TI, Tobih-Ojeanelo JI, Ramon-Yusuf HI, Olanrewaju A, Afuh RN, Adenikinju J, Amosu O, Yusuf A. Comprehensive review of current management guidelines of chronic kidney disease. Medicine (Baltimore). 2023 Jun 9;102(23):e33984. doi: 10.1097/MD.0000000000033984. PMID 37335639
- [Background] Chan SW. Chronic Disease Management, Self-Efficacy and Quality of Life. J Nurs Res. 2021 Feb 1;29(1):e129. doi: 10.1097/JNR.0000000000000422. No abstract available. PMID 33427791
- [Background] Halpin DMG, Criner GJ, Papi A, Singh D, Anzueto A, Martinez FJ, Agusti AA, Vogelmeier CF. Global Initiative for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease. The 2020 GOLD Science Committee Report on COVID-19 and Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2021 Jan 1;203(1):24-36. doi: 10.1164/rccm.202009-3533SO. PMID 33146552